CLINICAL TRIAL: NCT01927523
Title: Improving Life Chances of Disadvantaged Youth: Testing Best-Practice Academic vs. Non-Academic Supports Through a Large-Scale Randomized Control Trial in Chicago
Brief Title: Improving Life Chances of Disadvantaged Youth: Testing Best-Practice Academic vs. Non-Academic Supports
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Chicago (Other)
Collaborators: MacArthur Foundation (Other); U.S. Department of Justice (U.S. Federal Agency); Crown Family Philanthropies (Other); Edna McConnell Clark Foundation (Unknown); Youth Guidance (Unknown); Match Education (Other); Chicago Public Schools (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: SBS IRB13-0691; IRB13-0691 (Other: Social & Behavioral Sciences Institutional Review Board)
Record Dates: First submitted 2013-08-15; First posted 2013-08-22 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Youth Violence; Crime; Educational Achievement
Keywords: Youth violence; Crime; Educational achievement
MeSH Terms: interventions — heterologous prime boost COVID-19 vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control group (No Intervention): These youth will not receive the non-academic cognitive behavioral programming nor the intensive academic mathematics tutoring.
- BAM Group Therapy & Match Math Tutoring (Experimental): These youth will receive both the non-academic cognitive behavioral programming and the intensive academic mathematics tutoring.
  Interventions: Behavioral: BAM; Other: Match
- BAM Group Therapy (Experimental): These youth will receive the non-academic cognitive behavioral programming.
  Interventions: Behavioral: BAM
- Match Math Tutoring (Experimental): These youth will receive the intensive academic mathematics tutoring.
  Interventions: Other: Match

INTERVENTIONS:
Behavioral: BAM — BAM (Becoming a Man), a cognitive-behavioral group therapy intervention.
  Arms: BAM Group Therapy; BAM Group Therapy & Match Math Tutoring
Other: Match — An intensive math tutoring program.
  Arms: BAM Group Therapy & Match Math Tutoring; Match Math Tutoring

SUMMARY:
The purpose of this study is to learn more about the most cost-effective way to improve the long-term life outcomes of disadvantaged youth, by comparing best practice academic supports to best-practice non-academic supports, and learning more about whether investing in both simultaneously has synergistic (more than additive) effects.

DETAILED DESCRIPTION:
Our University of Chicago Crime Lab research team will carry out a 2 x 2 randomized experiment, in which some male youth are randomly assigned to receive what we believe to be best-practice intensive academic supports (high-dosage math tutoring provided by Match Education of Boston), or what we believe to be best-practice non-academic supports, for which we have identified Youth Guidance's Becoming a Man (BAM) program that provides a version of cognitive behavioral therapy (CBT), or to receive both, or neither (control condition).

The University of Chicago Education Lab research team will be carrying out a randomized controlled trial of this promising academic intervention during both the 2013-14 and 2014-15 academic years in partnership with the Chicago Public Schools (CPS) and Match Education.

The BAM intervention is a version of CBT adapted to help promote pro-social life outcomes among disadvantaged male youth. BAM includes in-school and after school programming designed to reduce overly-automatic behavior that can lead to problem outcomes, encourage youth to reflect on their decision-making heuristics, or promote meta-cognition (to "think about thinking"). By helping youth learn and practice new ways to manage their emotional responses to difficult situations through stories, role-playing, small group exercises, and homework, the program encourages what psychologists call "cognitive restructuring," designed to generate lasting gains in youths' behaviors. BAM is a program of Youth Guidance (YG), a Chicago-area non-profit that has been serving Chicago children for over 80 years, and currently provides services to thousands of students across more than 70 schools through a partnership with the Chicago Public Schools (CPS) that dates back more than four decades. YG will implement the BAM intervention during the 2013-15 academic years in some of the most distressed schools in Chicago's south and west sides.

The Match Tutors program expands on the nationally recognized innovation of high-dosage, in-school-day tutoring developed in the three Match Charter Public Schools in Boston. Tutoring is embedded into the school day as an elective class, as a supplement to the regular classroom math teacher. Every student works with a full-time, professional tutor in addition to their other classes, so that the class offered by Match Tutors will be given for credit, not as a pull-out or after school intervention As a regular part of their school day, students will attend tutoring for 50 minutes a day, 5 days a week. The tutoring course, entitled Mathematics Lab, has been granted credit-bearing status by CPS and will be offered each semester within a school year so that students will earn one elective credit upon completion of the course. Math Lab offers a standards-based curriculum that is individualized to each student's needs with the goal of complementing the work done in math classes - preparing students for city and state math assessments, enabling them to pass math class finals, and helping students build skills and habits of learning that will help them succeed in school and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Lowest-performing Chicago Public School high schools, based on dropout rate, scores on academic rating scale, and where fewer than 10% of students met state standards on the Prairie State Achievement Exam
* School administrators were enthusiastic about the program and agreed to terms and conditions of the experimental design
* Male youth within these schools who are rising 9th and 10th graders in AY (Academic Year) 2013-14 and 2014-15.

Exclusion Criteria:

* Youth who have missed >60% of days during AY2012-13 and AY2013-14 (through March), and so would not be expected to show up in school enough during intervention years (AY2013-15) to benefit from school-based programming
* Youth who have failed >75% of classes during AY2012-13 and AY2013-14 (through March)
* Youth who have IEP (Individualized Education Program) designations for autism, speech and language disabilities, "educable mentally handicapped", and traumatic brain injury

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5344 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in Violent Crime Arrests | 1-year, 2-year, 3-year, 4-year, 5-year
  Number of violent crime arrests, obtained from Chicago Police Department and Illinois State Police administrative databases
Change in other arrests (property, drug, and other) | 1-year, 2-year, 3-year, 4-year, 5-year
  Number of non-violent crime arrests, including property crimes, drug crimes, and other crimes, obtained from Chicago Police Department and Illinois State Police administrative databases
Change in index of CPS schooling outcomes | 1 year, 2 years, 3 years, 4 years
  Index of standardized (in Z-score form) outcomes for school persistence, absences, student misconducts, course grades

SECONDARY OUTCOMES:
Change in absentee Rate | 1-year, 2-year, 3-year, 4-year, 5-year
  Number of school absences, obtained from Chicago Public Schools administrative database
Change in Student Misconduct | 1-year, 2-year, 3-year, 4-year, 5-year
  Number of school misconduct infractions, obtained from Chicago Public Schools administrative database
Change in Total Courses Failed | 1-year, 2-year, 3-year, 4-year, 5-year
  Number of total school courses failed, obtained from Chicago Public Schools administrative database
Change in School persistence | 1 year, 2 years, 3 years, 4 years, 5 years
  Measure from CPS student records of school persistence (enrollment or graduation status by end of academic year).
Change in Math achievement | 2 years
  Performance on math standardized achievement test scores

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ludwig, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States